CLINICAL TRIAL: NCT03032354
Title: Effect of Lactobacillus Rhamnosus GG and Bifidobacterium Lactis BB 12 on Beta-cell Function in Children With Newly Diagnosed Type 1 Diabetes - a Randomized Controlled Trial
Brief Title: Probiotics in Newly Recognized Type 1 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Hanna Szajewska, Prof., Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AgaLidka
Record Dates: First submitted 2017-01-05; First posted 2017-01-26 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-01

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: probiotics; children; remission
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Probiotics; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics arm: Probiotics group (Experimental): combination of probiotics: Lactobacillus rhamnosus GG and Bifidobacterium lactis BB12 in the same capsule
  Interventions: Drug: Lactobacillus rhamnosus GG and Bifidobacterium lactis BB12
- Placebo arm: Placebo group (Placebo Comparator): Placebo - maltodextrin
  Interventions: Other: Placebo, (Placebo group)

INTERVENTIONS:
Drug: Lactobacillus rhamnosus GG and Bifidobacterium lactis BB12 — Combination therapy of probiotics during 6 months
  Other Names: Probiotics
  Arms: Probiotics arm: Probiotics group
Other: Placebo, (Placebo group) — Placebo during 6 months
  Other Names: Maltodextrin
  Arms: Placebo arm: Placebo group

SUMMARY:
They are major genera of bacteria that make up the colon flora in human, constitute intestinal microbial homeostasis, inhibit growth of pathogens, improve the gut mucosal barrier and modulate local and systemic immune responses. Changes in gut microbiota can influence the immune system by increasing gut permeability, intestinal inflammation, and impaired oral tolerance in type 1 diabetes.Taken together, the data imply that bacteriotherapy may potentially be used as a tool to modulate the immune system for preventing islet destruction. Supplementation of Lactobacillus rhamnosus GG and Bifidobacterium lactis BB12 improved blood glucose control in normoglycaemic pregnant women and reduced the frequency of gestational diabetes mellitus

Aim of the study:

The effect of Lactobacillus rhamnosus GG and Bifidobacterium lactis BB12 on beta-cell function in children with newly diagnosed type 1 diabetes: a randomized, double blind, placebo-controlled trial.

Primary end point:

Area under the curve (AUC) of c-peptide level during during fasting and at 30,60,90,120 min following the start of the meal

Intervention:

Included patients will be randomly assigned to receive a combination of Lactobacillus rhamnosus GG and Bifidobacterium lactis BB12 (Probiotics Group ) or placebo (Placebo Group ) during six months.

The expected results:

Beneficial effect of Lactobacillus rhamnosus GG and Bifidobacterium lactis BB12 on beta-cell function shown in the properly performed, methodologically accurate study would create a rationale for its routine use in patients with newly diagnosed type 1 diabetes.

DETAILED DESCRIPTION:
Intervention:

At the 6-month follow-up visit will be evaluated adherence and occurrence of side effects of the study procedure. The outcome measures will be assessed at the beginning of the study, and at the 6 and 12-month follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes confirmed by clinical history and the presence of at least one positive autoantibody: anti-glutamic acid decarboxylase (anti-GAD), islet antigen 2 (IA2), islet cell antibody ( ICA)
* Fasting c-peptide level >/= 0.4 ng/ml
* The diagnosis of diabetes during the last 60 days
* Consent to participate in the study

Exclusion Criteria:

* Antibiotic-therapy during last 4 weeks
* Taking of probiotics during last 2 weeks
* Intestinal infection during last 2 weeks
* Intestinal chronic diseases

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2017-07-15 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Area under the curve (AUC) during fasting and at 30,60,90,120 min following the start of the meal | 120 min responses to a mixed meal

SECONDARY OUTCOMES:
Insulin requirement (U / kg body mass ) | up 60 days from diabetes recognition, at 3th, 6th, 12th month
HbA1c | up to 60 days from diabetes recognition, at 3th, 6th, 12th month
Weight in kilograms | up to 60 days from diabetes recognition, and at 3th, 6th, 12th month
Number of participants with abnormal laboratory values and/or adverse events that are related to treatment ( eg.abdominal pain, diarrhea , constipation , vomiting,flatulence) | at 3th, 6th, 12th month
Occurrence of other autoimmune diseases | at 12th month
Height in meters | up to 60 days from diabetes recognition, and at 3th, 6th, 12th month
BMI in kg/m2 | up to 60 days from diabetes recognition, and at 3th, 6th, 12th month
BMI score | up to 60 days from diabetes recognition, and at 3th, 6th, 12th month
severe hypoglycemia | up to 60 days from diabetes recognition, at 3th, 6th, 12th month
ketoacidosis | up to 60 days from diabetes recognition, at 3th, 6th, 12th month
Fasting c- peptide concentrations in ng/ml | up to 60 days from diabetes recognition, and in: 6th, 12th month

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Szypowska, Assoc. Prof., Principal Investigator — Medical University of Warsaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kriegel MA, Sefik E, Hill JA, Wu HJ, Benoist C, Mathis D. Naturally transmitted segmented filamentous bacteria segregate with diabetes protection in nonobese diabetic mice. Proc Natl Acad Sci U S A. 2011 Jul 12;108(28):11548-53. doi: 10.1073/pnas.1108924108. Epub 2011 Jun 27. PMID 21709219
- [Background] Greenbaum CJ, Beam CA, Boulware D, Gitelman SE, Gottlieb PA, Herold KC, Lachin JM, McGee P, Palmer JP, Pescovitz MD, Krause-Steinrauf H, Skyler JS, Sosenko JM; Type 1 Diabetes TrialNet Study Group. Fall in C-peptide during first 2 years from diagnosis: evidence of at least two distinct phases from composite Type 1 Diabetes TrialNet data. Diabetes. 2012 Aug;61(8):2066-73. doi: 10.2337/db11-1538. Epub 2012 Jun 11. PMID 22688329
- [Background] Effect of intensive therapy on residual beta-cell function in patients with type 1 diabetes in the diabetes control and complications trial. A randomized, controlled trial. The Diabetes Control and Complications Trial Research Group. Ann Intern Med. 1998 Apr 1;128(7):517-23. doi: 10.7326/0003-4819-128-7-199804010-00001. PMID 9518395
- [Background] Shapiro AM, Ricordi C, Hering BJ, Auchincloss H, Lindblad R, Robertson RP, Secchi A, Brendel MD, Berney T, Brennan DC, Cagliero E, Alejandro R, Ryan EA, DiMercurio B, Morel P, Polonsky KS, Reems JA, Bretzel RG, Bertuzzi F, Froud T, Kandaswamy R, Sutherland DE, Eisenbarth G, Segal M, Preiksaitis J, Korbutt GS, Barton FB, Viviano L, Seyfert-Margolis V, Bluestone J, Lakey JR. International trial of the Edmonton protocol for islet transplantation. N Engl J Med. 2006 Sep 28;355(13):1318-30. doi: 10.1056/NEJMoa061267. PMID 17005949
- [Background] Laitinen K, Poussa T, Isolauri E; Nutrition, Allergy, Mucosal Immunology and Intestinal Microbiota Group. Probiotics and dietary counselling contribute to glucose regulation during and after pregnancy: a randomised controlled trial. Br J Nutr. 2009 Jun;101(11):1679-87. doi: 10.1017/S0007114508111461. Epub 2008 Nov 19. PMID 19017418
- [Background] Luoto R, Laitinen K, Nermes M, Isolauri E. Impact of maternal probiotic-supplemented dietary counselling on pregnancy outcome and prenatal and postnatal growth: a double-blind, placebo-controlled study. Br J Nutr. 2010 Jun;103(12):1792-9. doi: 10.1017/S0007114509993898. Epub 2010 Feb 4. PMID 20128938
- [Result] Badami E, Sorini C, Coccia M, Usuelli V, Molteni L, Bolla AM, Scavini M, Mariani A, King C, Bosi E, Falcone M. Defective differentiation of regulatory FoxP3+ T cells by small-intestinal dendritic cells in patients with type 1 diabetes. Diabetes. 2011 Aug;60(8):2120-4. doi: 10.2337/db10-1201. Epub 2011 Jun 6. PMID 21646390
- [Result] Hara N, Alkanani AK, Ir D, Robertson CE, Wagner BD, Frank DN, Zipris D. The role of the intestinal microbiota in type 1 diabetes. Clin Immunol. 2013 Feb;146(2):112-9. doi: 10.1016/j.clim.2012.12.001. Epub 2012 Dec 11. PMID 23314185
- [Result] Ludvigsson J, Faresjo M, Hjorth M, Axelsson S, Cheramy M, Pihl M, Vaarala O, Forsander G, Ivarsson S, Johansson C, Lindh A, Nilsson NO, Aman J, Ortqvist E, Zerhouni P, Casas R. GAD treatment and insulin secretion in recent-onset type 1 diabetes. N Engl J Med. 2008 Oct 30;359(18):1909-20. doi: 10.1056/NEJMoa0804328. Epub 2008 Oct 8. PMID 18843118
- [Result] American Diabetes Association. Standards of medical care in diabetes--2014. Diabetes Care. 2014 Jan;37 Suppl 1:S14-80. doi: 10.2337/dc14-S014. No abstract available. PMID 24357209
- [Result] Mejia-Leon ME, Petrosino JF, Ajami NJ, Dominguez-Bello MG, de la Barca AM. Fecal microbiota imbalance in Mexican children with type 1 diabetes. Sci Rep. 2014 Jan 22;4:3814. doi: 10.1038/srep03814. PMID 24448554
- [Result] Patelarou E, Girvalaki C, Brokalaki H, Patelarou A, Androulaki Z, Vardavas C. Current evidence on the associations of breastfeeding, infant formula, and cow's milk introduction with type 1 diabetes mellitus: a systematic review. Nutr Rev. 2012 Sep;70(9):509-19. doi: 10.1111/j.1753-4887.2012.00513.x. PMID 22946851
- [Result] Murri M, Leiva I, Gomez-Zumaquero JM, Tinahones FJ, Cardona F, Soriguer F, Queipo-Ortuno MI. Gut microbiota in children with type 1 diabetes differs from that in healthy children: a case-control study. BMC Med. 2013 Feb 21;11:46. doi: 10.1186/1741-7015-11-46. PMID 23433344
- [Result] Vaarala O. Human intestinal microbiota and type 1 diabetes. Curr Diab Rep. 2013 Oct;13(5):601-7. doi: 10.1007/s11892-013-0409-5. PMID 23934614
- [Result] Vaarala O, Atkinson MA, Neu J. The "perfect storm" for type 1 diabetes: the complex interplay between intestinal microbiota, gut permeability, and mucosal immunity. Diabetes. 2008 Oct;57(10):2555-62. doi: 10.2337/db08-0331. PMID 18820210
- [Result] de Goffau MC, Luopajarvi K, Knip M, Ilonen J, Ruohtula T, Harkonen T, Orivuori L, Hakala S, Welling GW, Harmsen HJ, Vaarala O. Fecal microbiota composition differs between children with beta-cell autoimmunity and those without. Diabetes. 2013 Apr;62(4):1238-44. doi: 10.2337/db12-0526. Epub 2012 Dec 28. PMID 23274889
- [Result] Hague A, Butt AJ, Paraskeva C. The role of butyrate in human colonic epithelial cells: an energy source or inducer of differentiation and apoptosis? Proc Nutr Soc. 1996 Nov;55(3):937-43. doi: 10.1079/pns19960090. No abstract available. PMID 9004335
- [Result] Peng L, Li ZR, Green RS, Holzman IR, Lin J. Butyrate enhances the intestinal barrier by facilitating tight junction assembly via activation of AMP-activated protein kinase in Caco-2 cell monolayers. J Nutr. 2009 Sep;139(9):1619-25. doi: 10.3945/jn.109.104638. Epub 2009 Jul 22. PMID 19625695
- [Result] Brown CT, Davis-Richardson AG, Giongo A, Gano KA, Crabb DB, Mukherjee N, Casella G, Drew JC, Ilonen J, Knip M, Hyoty H, Veijola R, Simell T, Simell O, Neu J, Wasserfall CH, Schatz D, Atkinson MA, Triplett EW. Gut microbiome metagenomics analysis suggests a functional model for the development of autoimmunity for type 1 diabetes. PLoS One. 2011;6(10):e25792. doi: 10.1371/journal.pone.0025792. Epub 2011 Oct 17. PMID 22043294
- [Result] Luopajarvi K, Savilahti E, Virtanen SM, Ilonen J, Knip M, Akerblom HK, Vaarala O. Enhanced levels of cow's milk antibodies in infancy in children who develop type 1 diabetes later in childhood. Pediatr Diabetes. 2008 Oct;9(5):434-41. doi: 10.1111/j.1399-5448.2008.00413.x. Epub 2008 May 21. PMID 18503496
- [Result] Turley SJ, Lee JW, Dutton-Swain N, Mathis D, Benoist C. Endocrine self and gut non-self intersect in the pancreatic lymph nodes. Proc Natl Acad Sci U S A. 2005 Dec 6;102(49):17729-33. doi: 10.1073/pnas.0509006102. Epub 2005 Nov 29. PMID 16317068
- [Result] Oikarinen M, Tauriainen S, Oikarinen S, Honkanen T, Collin P, Rantala I, Maki M, Kaukinen K, Hyoty H. Type 1 diabetes is associated with enterovirus infection in gut mucosa. Diabetes. 2012 Mar;61(3):687-91. doi: 10.2337/db11-1157. Epub 2012 Feb 7. PMID 22315304
- [Result] King C, Sarvetnick N. The incidence of type-1 diabetes in NOD mice is modulated by restricted flora not germ-free conditions. PLoS One. 2011 Feb 25;6(2):e17049. doi: 10.1371/journal.pone.0017049. PMID 21364875
- [Result] Roesch LF, Lorca GL, Casella G, Giongo A, Naranjo A, Pionzio AM, Li N, Mai V, Wasserfall CH, Schatz D, Atkinson MA, Neu J, Triplett EW. Culture-independent identification of gut bacteria correlated with the onset of diabetes in a rat model. ISME J. 2009 May;3(5):536-48. doi: 10.1038/ismej.2009.5. Epub 2009 Feb 19. PMID 19225551
- [Result] Valladares R, Sankar D, Li N, Williams E, Lai KK, Abdelgeliel AS, Gonzalez CF, Wasserfall CH, Larkin J, Schatz D, Atkinson MA, Triplett EW, Neu J, Lorca GL. Lactobacillus johnsonii N6.2 mitigates the development of type 1 diabetes in BB-DP rats. PLoS One. 2010 May 6;5(5):e10507. doi: 10.1371/journal.pone.0010507. PMID 20463897
- [Derived] Groele L, Szajewska H, Szalecki M, Swiderska J, Wysocka-Mincewicz M, Ochocinska A, Stelmaszczyk-Emmel A, Demkow U, Szypowska A. Lack of effect of Lactobacillus rhamnosus GG and Bifidobacterium lactis Bb12 on beta-cell function in children with newly diagnosed type 1 diabetes: a randomised controlled trial. BMJ Open Diabetes Res Care. 2021 Mar;9(1):e001523. doi: 10.1136/bmjdrc-2020-001523. PMID 33771763
- [Derived] Groele L, Szajewska H, Szypowska A. Effects of Lactobacillus rhamnosus GG and Bifidobacterium lactis Bb12 on beta-cell function in children with newly diagnosed type 1 diabetes: protocol of a randomised controlled trial. BMJ Open. 2017 Oct 11;7(10):e017178. doi: 10.1136/bmjopen-2017-017178. PMID 29025837